CLINICAL TRIAL: NCT02935920
Title: A Study on Optimizing Follow-up for Postmenopausal Women With Breast Cancer Treated With Adjuvant Endocrine Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OOBS
Record Dates: First submitted 2016-08-03; First posted 2016-10-18 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: PRO, follow up
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual, tailored follow-up (Experimental): Patient symptoms are evaluated by the use of PRO-data to uncover the needs of a consultation. The outcome of the questionnaire is used to customize the follow-up program to the individual patient.
  Interventions: Behavioral: Individualized, tailored follow-up program
- Standard follow-up (No Intervention): Scheduled clinical examination every six months throughout the course of adjuvant treatment. Performed by a doctor or nurse.

INTERVENTIONS:
Behavioral: Individualized, tailored follow-up program — Individualized follow-up in the context of shared decision making, with the use of PRO-data to evaluate the patient needs of consultations.
  Arms: Individual, tailored follow-up

SUMMARY:
Background:

In February 2015 the Danish Health and Medicines Authority published new clinical guidelines describing how cancer patients should be followed. It is recommended that patients receiving specific oncological treatment such as endocrine therapy be followed at the department of oncology responsible for the treatment and providing the medication. There is no evidence that routine examinations improve overall survival after breast cancer. Mammography is the only specific examination to be offered to asymptomatic women after treatment for breast cancer

Aims of the study:

The hypothesis is that individualized follow-up with the introduction of Patient Reported Outcome (PRO) data will help postmenopausal women regain control of health related self-care and encourage them to a larger extent to take part in their follow-up after cancer treatment. This is believed to improve the health related quality of life and increase the positive experience of the follow-up program.

Design:

Patients are randomly assigned to the department's standard control program or an individualized solution in the context of shared decision making. PRO data will be used to evaluate the patient's need for consultations.

Primary outcome:

Evaluation of the experience and feasibility of PRO data in connection with individualized follow-up of postmenopausal women with breast cancer. Systematically applying PRO data we will uncover patient needs, empower the patients to take part in shared decision making, and improve the current follow-up in the sense of a more patient-centered care and tailored follow-up.

DETAILED DESCRIPTION:
Introduction

The purpose of the present follow-up program, after treatment for early stage breast cancer, is to detect local and systemic recurrences, new primary tumors in the breasts, and secondary cancer. Furthermore, the clinicians aim to provide the patients with social and psychological support, if needed, and support them in managing side effects to their primary treatment and current endocrine therapy.

Patient reported outcomes (PRO)

It has been demonstrated that clinicians systematically underestimate patient symptoms, and that many symptoms go unrecognized. Patients frequently deal with symptoms of both physical and psychological origin between visits and may have been carrying them for an unacceptable period of time, because of the natural thresholds for calling the department. Also, they may forget to communicate the symptoms at their appointment in the clinic. If the symptoms persist and are revealed at the consultation, they are commonly more severe to the patient at this time than when they first appeared.

Information about the patient's individual symptoms and health status during cancer treatment and follow-up is currently obtained by the clinician as part of the communication with the patient. This approach is not systematic and cannot be used to monitor symptoms development over time. However, knowledge of health status is essential for assessing and improving well-being and rehabilitation in cancer care aiming the best possible outcome. Fewer symptoms may thus be an indication of whether supportive care has been effective, while the appearance of new symptoms may reflect recurrence in an early stage. Electronic registration of systemically obtained PRO data in clinical practice can be a method to improve the quality of the follow-up program .

PRO data is information about patient experienced symptoms, functional capacity, and quality of life and has not yet been implemented as a systemically obtained measurement in the follow-up program. According to the US Food and Drug Administration (FDA) PRO data is: "any report of the status of a patient's health condition that comes directly from the patient, without interpretation of the patient's response by a clinician or anyone else". PRO data are typically collected through a questionnaire in which measurements are repeated over time. This allows continuous monitoring of the patient health status. PRO data is a tool to improve healthcare quality and the key to organize and deliver healthcare in a way beneficial to the patients. Today, PRO data are not routinely obtained during follow-up, but the new guidelines from the Danish Health and Medicines Authority recommend the use of PRO data. The implementation faces several challenges due to the extra effort by the staff, the development of appropriate electronic equipment, and determination of the proper use in different parts of the healthcare system.

Providing information congruent with patient needs is important to denote patient involvement and satisfaction, and it may also affect the health-related quality of life. Shared decision making is one of the most recent models fostered by healthcare research and aims to establish a partnership between the healthcare professional and the patient. The model describes how decisions should be made. It is centered on the idea that the healthcare professional communicates medical knowledge to the patient, and that the patient's perspectives, preferences and rights are included in the clinical conversation. The exchange of knowledge and information is one of the most important preconditions to carry out shared decision making in clinical practice.

The study is a randomized trial in which patients are assigned to the department's standard follow-up program or to individualized follow-up in the context of shared decision making with PRO-data guiding the clinician as to the patient's need for consultations in the clinic by a nurse, doctor, physiotherapist, social workers and/or psychologist. The individual follow-up program also offers the possibility of consulting a sexologist and a coach, probably with an extent of self-payment. In both programs the patients can call the department and make arrangement for an urgent appointment. Only the individualized program offers email consultation and patient influence as to how much effort they want to spend on their follow-up.

Data collection:

PRO data will be handled electronically in the software program SurveyXact, where the patients obtain access to different questionnaires through secured links.

The clinicians and nurses who take care of the patients in either of the programs are requested to fill out a brief questionnaire after seeing each patient to register the complaints or concerns that led to the contact, and what was to solve the problem. In compliance with departmental guidelines, the patients will be recommended supportive medical care, referred to physiotherapy, plastic surgery, or extraordinary imaging.

The patients in both programs are also requested to fill out a patient satisfaction questionnaire after each consultation and a CollaboRATE questionnaire containing three brief questions to measure the level of shared decision making.

Perspectives:

The socioeconomic aspects related to the introduction of a patient centered, individualized follow-up program, where resources are spent on those in need of them, are of great importance in the Danish healthcare system. The results of this study can be used nationally in providing tailored follow-up to this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal at the time of diagnosis (menostasis > 12 months. Bilateral salpingo-oophorectomy)
* Complete disease remission after primary operation
* Histologically confirmed hormone-receptor positive breast cancer, 1% or more of the tumor cells express hormone receptors
* High-risk profile with a 10-year recurrence of more than 10%
* Planned adjuvant endocrine therapy regardless of other adjuvant therapy to be initiated within 1 month or initiated within the last 9 months.
* Written and verbally informed consent
* Able to read and speak Danish
* Access to a computer and an email-account

Exclusion Criteria:

* Patient followed regularly as part of a research protocol
* Women postmenopausal due to surgery on the ovaries/uterus age < 50
* Prognostic low grade risk of recurrence (tumor size 10 mm or less, lymph node negative, ductal carcinoma grade 1 and lobular carcinoma grade 1 or 2)

Ages: 45 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
The difference in PREM (patient reported experience measure) as reported by patients in the individualized and standard follow-up groups, respectively | 2 years
  Every three months the patients in both groups are requested to fill out a patient satisfaction questionnaire (PEQ) concerning their follow-up program. A single item with scores between 1 and 5 will be used to evaluate the difference between the 2 groups (1 is very satisfied and 5 is very dissatisfied)

SECONDARY OUTCOMES:
Comparison of resources spent on individualized follow-up based on PRO-data and standard follow-up. | 2 years
  On a yearly basis the two programs will be compared as to number of consultations, telephone calls, and e-mail consultations per patient, including time spent on zoledronic acid infusion and evaluation of PRO questionnaires. Data are obtained from the medical journals.
The difference in CollaboRATE-score between the individualized and standard follow-up. | 2 years
  The CollaboRATE questionnaire contains three brief questions to measure the level of patient involvement and shared decision-making.
Comparison of Health related quality of life in the individualized follow-up versus standard follow-up. | 2 years
  Health related quality of life evaluated by comparison of the global score of the quality of life questionnaire EORTC QLQ C-30, which patients are asked to fill out every three months.
Elucidation of issues of importance and concern to postmenopausal woman with breast cancer in adjuvant endocrine therapy during follow-up after primary treatment. What symptoms and side effects trouble them most during follow-up? | 2 years
  The nurse or clinician places the main concern/complaint leading to the consultation into one of five categories; 1) Sign of or worry about recurrence or a new tumor, 2) Side effects to the endocrine treatment, 3) Side effects to the primary treatment. 4) Psychosocial problems, 5) Other. The differences in complaints between the standard and individualized follow-up programs will then be described.
Evaluation of current information level during primary treatment | 2 years
  How do patients experience the given information? The demographic questionnaire at baseline will elucidate the patient's current level of insight into her disease. Does she feel knowledgeable enough about her situation and options? Has she searched for information elsewhere or would she rather not know too many details?

CONTACTS AND LOCATIONS:
Overall Officials: Karina D. Steffensen, MD, PhD, Study Chair — Vejle Hospital; Cathrine L. Riis, MD, Principal Investigator — Vejle Hospital
Locations (1):
- Vejle hospital, Department of Oncology, Vejle, Region of Southen Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No